CLINICAL TRIAL: NCT06640153
Title: Preoperative Evaluation of Resectability in Gastroesophageal Junction and Upper Gastric Adenocarcinoma Utilizing Multi-Parametric MRI and CT Imaging.
Brief Title: MRI and CT in Gastroesophageal Junction or Upper Gastric Adenocarcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-587
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer, Gastroesophageal Junction Cancer
Keywords: MR; CT; Adenocarcinoma of the Gastroesophageal Junction; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Gastroesophageal junction or upper gastric adenocarcinoma: Patients with biopsy verified gastroesophageal junction or upper gastric adenocarcinoma undergo mpMRI in addition to conventional CT imaging
  Interventions: Diagnostic Test: mpMRI

INTERVENTIONS:
Diagnostic Test: mpMRI — Gastroesophageal junction or upper gastric adenocarcinoma patients undergo mpMRI at siewert classification, length of esophageal involvement, primary staging and restaging

SUMMARY:
Accurate preoperative Siewert classification, precise assessment of the extent of esophageal involvement, and staging is crucial for determining the appropriate surgical approach and achieving negative resection margins. The purpose of this study is to investigate the diagnostic performance of the Multi-parametric magnetic resonance imaging (mpMRI) and computed tomography (CT) in gastroesophageal junction and upper gastric cancers.

DETAILED DESCRIPTION:
Despite a continuous decline in the incidence of gastric cancer in recent years, the morbidity and mortality rates associated with the gastroesophageal junction and upper gastric cancers remain elevated. Consequently, it is imperative to develop more refined and individualized precision strategies for screening, diagnosis, surgical intervention, and comprehensive treatment. Due to the unique anatomical location, considerable debate exists regarding the critical aspects of its surgical management in clinical practice. Multiparametric MRI offers significant anatomical benefits due to its high soft tissue resolution, and its functional imaging capabilities present promising applications. With advancements in abdominal imaging technology, novel techniques such as high-order diffusion imaging and compressed sensing technology have facilitated high-resolution MRI of the stomach during free breathing, which is now implemented in clinical practice. Prior research has demonstrated that individualized gastric MRI scanning consistently yields superior image quality, and MRI provides greater accuracy than CT in preoperative staging assessments. Nonetheless, the comparative study of MRI and CT in patients with gastroesophageal junction and upper gastric cancers remains to be elucidated.

ELIGIBILITY:
Inclusion Criteria:

1. patients with gastric cancer confirmed by preoperative gastroscopic biopsy;
2. underwent standardized mpMRI and CT examination;
3. patients with complete postoperative pathological data and pathological results of gastroesophageal Junction or upper gastric adenocarcinoma;

Exclusion Criteria:

1. combined with other tumors;
2. Clinical and imaging data were missing or could not meet the research needs;
3. the location of lesions could not be determined;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gastroesophageal junction or upper gastric adenocarcinoma who are candidates for radical surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-08-24 (Estimated); Study Completion 2027-08-24 (Estimated)

PRIMARY OUTCOMES:
Siewert classification | 2 years
  Compare the findings of multiparametric MRI and CT in the Siewert classification (Types I, II, and III) against a histopathological reference standard, evaluating sensitivity, specificity, positive predictive value, and negative predictive value.
length of esophageal involvement | 2 years
  The accuracy and AUC of length of esophageal involvement (not involved, 0-2cm, 2-3cm, 3-4cm, >4cm) evaluated by CT and MRI.
Staging | 2 years
  Compare the cancer stage (according to AJCC 8th edition TNM-classification) as determined by mpMRI compared to CT at primary staging and at restaging. The proportion of upgraded, downgraded, and right patients are determined.

SECONDARY OUTCOMES:
Survival time and recurrence time | 3 years
  3-year overall survival
  1-year and 3-year recurrence free survival
The number of patients with complications | Within 30 days after the day of operation
  The morbidity and mortality rates within 30 days after the day of operation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT06640153/ICF_000.pdf